CLINICAL TRIAL: NCT00769210
Title: The Effect of Simvastatin Therapy on the Expression of Procoagulant and Inflammatory Markers in Heart Failure
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, mark munger, Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012064; IRB# 00013639
Record Dates: First submitted 2007-12-22; First posted 2008-10-09 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40 mg tablet
  Other Names: Zocor

SUMMARY:
Our proposed research will examine whether treatment with simvastatin alters expression and activity of monocyte TF, whether polymorphisms in the TF gene alter the therapeutic effect and what effect treatment has on inflammatory markers in heart failure. The results of this study may assist in tailoring statin therapy to specific characteristics, such as inflammatory state, of heart failure patients. If treatment with simvastatin significantly lowers TF expression, this may reduce the risk of thromboembolic events in patients with heart failure, thus reducing mortality and morbidity. If the treatment effect varies based on the TF genotype, this may define an identifiable population in whom statin therapy may be more beneficial than the population as a whole.

DETAILED DESCRIPTION:
Heart failure is a significant public health problem in the United States. There are more than five million heart failure patients in America and this number grows by over 550,000 new cases each year.1 Heart failure is the primary diagnosis for nearly one million hospital admissions each year and another two million patients are admitted with a secondary diagnosis of heart failure, making it the single largest expense for Medicare.1 Furthermore, heart failure causes or contributes to more than 300,000 deaths each year and, in spite of advances in treatment, 70-80% of patients with heart failure will die within 8 years.1, 2 Therefore, heart failure is one of, if not the most important socioeconomic health problems of the 21st century.

Heart failure patients are at increased risks for thromboembolic events. Autopsy results from heart failure patients report a 50% to 60% incidence of thromboembolic events.3-5 Besides known thromboembolic risk factors associated with the heart failure state (such as blood stasis in a poorly contracting left ventricle, endothelial dysfunction and neuroendocrine activation), elevated TF expression may also contribute to enhanced thromboembolic risk. Recent evidence from our laboratory shows that functional TF procoagulant activity (TF-PCA) in monocytes is increased significantly by 2.8-fold in heart failure patients (n=48) compared to healthy controls (n=25) (p=0.03) (Figure 1), while the natural inhibitor tissue factor pathway inhibitor (TFPI) showed no significant difference.6 The heart failure subjects were subsequently followed to death, transplant, or clinical event (i.e. heart failure hospitalization, arrhythmia, acute coronary event, thromboembolic event, death or cardiac transplant). When TF-PCA values were divided at the median, the upper 50-percentile demonstrated a trend toward increased mortality (p=0.06) with a significant increase in clinical events (p=0.04) compared to the lower 50-percentile (Figure 2).

Elevated TF expression is believed to play an integral role in intravascular coagulation seen in coronary artery disease.7-9 Human atherosclerotic plaques are highly thrombogenic, and exhibit high levels of TF antigen and functional TF procoagulant activity.10-15 In addition, TF antigen is higher in plaques from patients with myocardial infarction and unstable angina than in those with stable angina.15 Recent evidence also shows that local TF inhibition by TFPI decreases the thrombogenicity of disrupted human atherosclerotic plaques.16 These data support that increased TF expression may mediate an increased risk of thromboembolic events.

Simvastatin, an antilipidemic agent of the HMG-CoA reductase inhibitor type, has been shown to decrease monocyte TF expression in vitro and ex vivo.17-20 In monocytes collected from both healthy volunteers and hyperlipidemic patients and stimulated with LPS (a potent inducer of TF) in vitro, simvastatin inhibits monocyte TF expression in a dose-dependent manner.17 In an in vivo model, hyperlipidemic patients receiving simvastatin exhibited a significant decrease in TF-Ag and TF-PCA from baseline (mean reduction 68% and 61%, respectively), while these TF parameters remained unchanged in the placebo group (p=0.0002).18 Whether simvastatin also decreases TF expression in heart failure is unknown.

Clinical studies of simvastatin and other statins have mostly been confined to their lipid-lowering effects. However, evidence also suggests that they improve outcomes in heart failure. In a post-hoc analysis of the Scandinavian Simvastatin Survival Study (4S), simvastatin 20-40 mg daily in patients with coronary heart disease significantly reduced the occurrence of heart failure (relative risk reduction 21.7%, p<0.015) and heart failure mortality (relative risk reduction 37%, p=0.014).21 Simvastatin also showed a non-significant trend in decreasing heart failure hospitalizations. An analysis of data from the PRAISE trial showed a 62% decrease in the risk of death in patients treated with statins, independent of their on-treatment cholesterol levels.22 The OMPTIMAAL trial also showed an improvement in survival of heart failure patients with statin therapy.23 In a cohort study by Horwich et al, statin use was associated with a reduction in the risk of heart transplant or death, again without regard to cholesterol levels.24 These results suggest that treatment with HMG-CoA reductase inhibitors have a beneficial effect, beyond that which would be expected from their ability to alter plasma lipid levels.

Two distinct common alleles of the tissue factor gene, designated - 1208 D and - 1208 I, have been identified.25 The two haplotypes had roughly equal frequencies in a sample of 2354 individuals.25 There are conflicting data on the effect of the alleles on TF expression, with one study showing lowered plasma TF and a decreased risk of venous thrombosis when the - 1208 D haplotype is present.25 Other studies have shown that the presence of the - 1208 D haplotype results in higher cellular expression of TF.26, 27 The effect of polymorphisms on the efficacy of statins in lowering TF is unknown, as are their clinical impact in heart failure.

A number of pro-inflammatory cytokines are elevated in heart failure. Evidence from our laboratory showed that Interleukin-6 (IL-6) levels were 75 pg/mL in NYHA class II-IV heart failure patients, compared to 0.4 pg/mL in healthy volunteers (p=0.002).28 Others have found similar elevations and have shown elevated IL-6 concentrations to be an independent predictor of worsening heart failure and adverse events.29-34 Statins have been shown to decrease expression of IL-6 in vitro, in coronary artery disease patients and in diabetes.35-40 Other inflammatory cytokines, such as IL-1/10 ratio and tissue necrosis factor (TNF), have also been implicated in procoagulant states and are potential targets of statin therapy.29, 31, 33 What effect statins have on the elevation of IL-6 and other cytokines in heart failure and what impact reduction of them with statins has on outcomes is unknown.

Our proposed research will examine whether treatment with simvastatin alters expression and activity of monocyte TF, whether polymorphisms in the TF gene alter the therapeutic effect and what effect treatment has on inflammatory markers in heart failure. The results of this study may assist in tailoring statin therapy to specific characteristics, such as inflammatory state, of heart failure patients. If treatment with simvastatin significantly lowers TF expression, this may reduce the risk of thromboembolic events in patients with heart failure, thus reducing mortality and morbidity. If the treatment effect varies based on the TF genotype, this may define an identifiable population in whom statin therapy may be more beneficial than the population as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 85 years
* Symptomatic heart failure, NYHA class I to III
* Left ventricular ejection fraction < 0.40
* Give written informed consent

Exclusion Criteria:

* Pregnant or lactating women. Women in reproductive years must have an active form of contraception (oral contraceptives, IUD, diaphragm, condoms or surgical sterilization) and a negative pregnancy test at study entry.
* Heart failure as the results of any of the following conditions:

  1. active myocarditis
  2. congenital heart disease
  3. uncorrected, hemodynamically significant stenotic valvular disease
  4. NYHA functional class IV symptoms
  5. Current or previous treatment with a statin Patients with plasma LDL-C concentrations higher than 130 mg/dL and any of the following conditions
  6. Ischemic cardiomyopathy
  7. Previous cardiovascular event (CVA, ACS event)
  8. Known coronary artery disease
  9. Unstable angina
* Presence of any progressive systemic disease that would be expected to impact the patient's outcome over the time course of the study
* Uncorrected endocrine disorders including primary aldosteronism, pheochromocytoma, hyperthyroidism, hypothyroidism, brittle type 1 diabetes mellitus
* Inherited disorders of lipid metabolism
* Evidence of significant renal disease (serum creatinine > 2.5 mg/dl), or hepatic disease (transaminase levels > three fold higher than laboratory normal)
* Inability or unwillingness to cooperate with study or give written informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Measure the effect of simvastatin treatment on the expression and activity of TF in patients with heart failure. | May 2005-June 2008

SECONDARY OUTCOMES:
Determine if polymorphisms in the gene coding for TF affect the impact of simvastatin therapy on tissue factor expression | May 2005-June 2008

CONTACTS AND LOCATIONS:
Overall Officials: Mark Munger, PharmD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States